CLINICAL TRIAL: NCT01038947
Title: A Cohort Dose-Escalation Phase 1 Study of Intramuscular Injection of Uricase-PEG 20
Brief Title: Safety and Efficacy Study of Intramuscular Uricase-PEG 20
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: EnzymeRx (Industry)
Responsible Party: Anthony Fiorino, MD, PhD, EnzymeRx, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENZ-102
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Uricase-PEG 20 (Experimental): Cohorts will receive ascending doses of Uricase-PEG 20 in a sequential manner. The study will enroll both single dose cohorts and multi-dose cohorts.
  Interventions: Biological: Uricase-PEG 20

INTERVENTIONS:
Biological: Uricase-PEG 20 — Intramuscular injection of Uricase-PEG 20 without premedication

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetics and pharmacodynamics of single and multiple intramuscular doses of Uricase-PEG 20

DETAILED DESCRIPTION:
Uricase is an enzyme (found in most mammals but not humans) that converts poorly soluble uric acid into highly soluble allantoin. Because humans lack uricase, they are prone to develop elevated levels of uric acid, which can form crystals in the joints and soft tissues. In those which chronically elevated uric acid, gout may develop. In the setting of acute rises in uric acid, seen for example in tumor lysis syndrome, uric acid crystals can damage the renal tubules. Uricase-PEG 20 is a recombinant uricase conjugated with multiple PEG molecules designed to prolong the half-life and decrease the immunogenicity of uricase. This study will characterize the safety, pharmacokinetics and pharmacodynamics of intramuscular Uricase-PEG 20, the anticipated route of administration to be used in future clinical development in gout.

ELIGIBILITY:
Inclusion Criteria:

* Serum uric acid > 6 mg/dL (men) or > 5 mg/dL (women)
* Clinical laboratory values within normal limits or not clinically significant
* Women should be menopausal or peri-menopausal

Exclusion Criteria:

* Prior exposure to uricase
* History of severe allergic reactions, or any allergy to PEG or pegylated products
* G6PD or catalase deficiency
* Medical condition that may interfere with ability to complete the study (e.g., uncontrolled diabetes or hypertension, congestive heart failure NYHA Class III or IV, history of myocardial infarction, immunosuppression, pregnancy)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-04 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Safety (assessment of signs and symptoms and clinical laboratory measurements following administration of Uricase-PEG 20, graded according to the Common Toxicity Criteria for Rheumatology, version 2.0) | Up to 35 days after dosing

SECONDARY OUTCOMES:
Pharmacokinetics (Uricase-PEG 20 serum concentration) | Up to 35 days after dosing
Pharmacodynamics (plasma uric acid concentration) | Up to 35 days after dosing
Immunogenicity | Up to 35 days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Anthony S Fiorino, MD, PhD, Study Director — EnzymeRx, LLC; Patricia Pardo, MD, Principal Investigator — MRA Clinical Research
Locations (2):
- United States (2):
  - MRA Clinical Research, Miami, Florida
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania

REFERENCES:
- [Background] Bomalaski JS, Holtsberg FW, Ensor CM, Clark MA. Uricase formulated with polyethylene glycol (uricase-PEG 20): biochemical rationale and preclinical studies. J Rheumatol. 2002 Sep;29(9):1942-9. PMID 12233890